CLINICAL TRIAL: NCT02021383
Title: "Lose 2 Win" Contests: A Novel Method to Motivate Weight Loss Maintenance Among College Students
Brief Title: Lose 2 Win A Novel Method to Motivate Weight Loss Maintenance Among College Students
Acronym: L2W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1207S16661; 20807 (Other Grant/Funding Number: UMN - Clinical and Translational Science Institute)
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Overweight; Obese
Keywords: Weight loss; Weight maintenance; Contingency Management; College students; Financial incentives
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Contest Plus (Experimental): The Contest Plus group were eligible to receive the financial incentives for weight loss maintenance at three monthly follow ups; weeks 16, 20 and 24. Eligible participants completed online surveys and in person weigh ins verifying weight maintenance. In addition to the financial incentives, participants in this group had bi-weekly in person meetings with a Registered Dietician during phase 2 (week 16-24) of the trial. They also received an in home scale to monitor weight daily.
  Interventions: Behavioral: Bi-weekly in person meetings with a Registered Dietician; Behavioral: Financial incentives for weight loss maintenance
- Control (No Intervention): The Control condition did not receive any intervention and were not eligible to win the lottery based incentive. Participants completed follow surveys (weeks 16, 20 and 24) and received remuneration for completing surveys and in person weigh in.
- Contest Only (Experimental): The Contest only group were eligible to receive the financial incentives for weight loss maintenance for maintaining weight lost at three monthly follow ups; weeks 16, 20 and 24. Eligible participants completed online surveys and in person weigh ins verifying weight maintenance.
  Interventions: Behavioral: Financial incentives for weight loss maintenance

INTERVENTIONS:
Behavioral: Bi-weekly in person meetings with a Registered Dietician — Participants in the Contest Plus group had the opportunity to receive 5 in person meetings with a Registered Dietician. These meetings took place bi-weekly and gave the participants a chance to discuss food consumption, physical activity, meal planning and assessed the participant's weight at each visit.
  Participants in the Contest only and Control group were not eligible to receive these meetings.
  Arms: Contest Plus
Behavioral: Financial incentives for weight loss maintenance — Participants in the Contest Plus and Contest Only groups were eligible for a lottery based financial incentive for maintaining their weight lost during phase 1 (Baseline to week 10) of the trial. There were three, month-long follow up assessments (weeks 16, 20 and 24) that participants were eligible for. The lottery prize was contingent upon the length of time they maintained their weight loss.
  Arms: Contest Only; Contest Plus

SUMMARY:
Investigators are conducting a randomized controlled trial with overweight and obese college students on the University of Minnesota campus. The primary outcome will be weight loss measured 12 months after study enrollment (corresponds to 10 months after the end of treatment).

DETAILED DESCRIPTION:
Approximately 30% of college students are overweight or obese. Intervening on excess weight early may eliminate obesity-related morbidity. Evidence supports use of monetary incentives to encourage weight-loss; questions remain about the efficacy of contingency management on weight loss maintenance.

"Lose 2 Win" contests in which participants who achieve weight-loss goals are eligible for cash prizes, appear well-suited for implementation on campuses. Our objective in this two-phase trial is to evaluate the feasibility, acceptability and efficacy of Lose 2 Win for weight-loss maintenance among college students.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years of age
* University of Minnesota Freshman, Sophomore, or Junior
* Plan on enrolling at the U of Minnesota through Spring 2013
* BMI greater than or equal to 26 and less than or equal to 35.5
* Have working internet and phone access
* Ability to read/write English
* Ability to safely engage in exercise

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Prior or planned weight loss surgery
* Having a special diet or being a member of an "organized weight loss program"
* Diagnosis of Diabetes
* Have had Binge Eating Disorder
* Have lost greater than or equal to 10 pounds in the last 3 months

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Maintenance of the weight lost from Baseline to Week 10 (Phase 1) measured ten months (week 52) after end of treatment (week 10). | Baseline, Week 10, Week 24, Week 52

SECONDARY OUTCOMES:
Change in physical activity from baseline on the Physical Activity Questionnaire at week 24 | Baseline, Week 24
Change in physical activity from baseline on the Physical Activity Questionnaire at week 52 | Baseline, Week 52
Change in nutritional quality of diet from baseline on the Block Food Questionnaire at week 24 | Baseline, Week 24
Change in nutritional quality of diet from baseline on the Block Food Questionnaire at week 52 | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Thomas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States